CLINICAL TRIAL: NCT06371911
Title: Benefit of Adding Cureety TechCare Telemonitoring to Usual Care During Injectable Anticancer Treatment: a Multicentric French Prospective Randomized Study: The OPTIMACURE Protocol
Brief Title: Benefit of Adding Cureety TechCare Telemonitoring to Usual Care During Injectable Anticancer Treatment
Acronym: OPTIMACURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Cureety (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-A02762-43
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-08

CONDITIONS: Adult Patients Initiating Injectable Anticancer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cureety telemonitoring (Experimental): The digital telemonitoring platform, Cureety, has been designed to facilitate the monitoring of signs and symptoms of treatment-specific AEs and disease progression. The platform integrates Cureety TechCare, a CE marked algorithm that is a class I medical device
  Interventions: Other: Cureety telemonitoring
- OPTIMA or equivalent programs (Active Comparator): The programs consist of three stages:
  1. The medical team make structured telephone calls with patients 2 to 3 days before the planned administration of injectable treatment. Adverse events and other relevant data are collected.
  2. Patients undergo biological tests within 48 hours of the appointment and the results are sent by the laboratory to the centre.
  3. Then, the physician assesses the data and decides whether to anticipate and validate the prescription of injectable treatments.
  Interventions: Other: OPTIMA or equivalent programs

INTERVENTIONS:
Other: Cureety telemonitoring — The digital telemonitoring platform, Cureety, has been designed to facilitate the monitoring of signs and symptoms of treatment-specific AEs and disease progression. The platform integrates Cureety TechCare, a CE marked algorithm that is a class I medical device
  Arms: Cureety telemonitoring
Other: OPTIMA or equivalent programs — The programs consist of three stages:
  1. The medical team make structured telephone calls with patients 2 to 3 days before the planned administration of injectable treatment. Adverse events and other relevant data are collected.
  2. Patients undergo biological tests within 48 hours of the appointment and the results are sent by the laboratory to the centre.
  3. Then, the physician assesses the data and decides whether to anticipate and validate the prescription of injectable treatments.
  Arms: OPTIMA or equivalent programs

SUMMARY:
Currently, during usual care, it is critical to assess whether a patient is apt to receive injectable anticancer treatment in the days prior to the administration. To assess this, blood tests are usually performed in the days leading up to the planned administration. A hospital staff member then telephones the patients and evaluates, using the tests results and other patient data (including the presence of adverse events (AEs) and Eastern Cooperative Oncology Group [ECOG] performance status), whether the patient is apt for treatment or whether the treatment needs to be deferred.

In France, the Centre François Baclesse in Caen (France) launched the OPTIMA program to optimize the prescription and preparation of chemotherapy in the ambulatory unit of the hospital.

A prospective study validating the OPTIMA program found that the prescription of chemotherapy was accurate with significantly reduced waiting times for patients between the planned appointment time and initiation of chemotherapyThe OPTIMA program is now part of usual care at the Centre François Baclesse.

Following the positive impact of both the OPTIMA and "Star" programs, several French healthcare centers have implemented similar programs. However, a large proportion of the data during the program are collected by telephone, particularly outgoing calls (from the hospital staff to patients). Thus, implementing these programs is expected to increase the number and/or duration of outgoing calls and consequently the workload of hospital staff.

Since the deployment of the OPTIMA program (between 2014 and 2016), and other equivalent programs, more and more patients have asked for the telephone calls to be replaced by a web-based application. Indeed, patients do not always respond to the telephone calls made by hospital staff, thus forcing staff to repeat calls several times. Also, some patients with language or hearing difficulties are unable to answer the questionnaires by telephone: a web-based alternative would be more appropriate for these patients.

Telemonitoring can collect blood test results and other patient data required to evaluate whether patients are apt for injectable cancer treatment. Telemonitoring can then identify the few patients that need to be contacted by hospital staff, thus reducing the number of outgoing telephone calls.

There is growing evidence of the benefits of adding telemonitoring to usual care for patients undergoing cancer treatment. The benefits include the early detection of AEs, improved quality of life (QoL), fewer admissions to emergency rooms or hospitalization, the longer remaining on chemotherapy for patients, and extended overall survival.

Cureety is a digital telemonitoring platform, specifically designed to monitor signs and symptoms of disease progression and AEs in cancer patients. The digital tool includes questionnaires for each class of medication to monitor patients' adverse events remotely. The data collected include blood results, treatment-related data (including delays, dose reductions), as well as QoL and safety data. In terms of safety, patients respond to an electronic patient-reported outcome (ePRO) questionnaire based on the NCI-CTCAE version (v)5.0. Depending on the responses, the Cureety TechCare algorithm classifies the patient state as "correct", "compromised", "to be monitored", or "critical". The patients are then notified of the actions to be taken according to their classification. In preparation for injectable cancer treatment, Cureety can collect the data necessary to evaluate whether patients are apt for treatment administration. The collection and evaluation of this data is expected to decrease outgoing calls by between 30% to 50%.

This study was designed to evaluate whether adding Cureety telemonitoring to usual care would reduce the number of outgoing calls for hospital staff during the management of patients undergoing injectable at one of the participating centers compared with the usual care including a program for anticipation of injectable treatment (OPTIMA program or equivalent).

ELIGIBILITY:
Inclusion criteria

* Patients that have provided written informed consent for study participation before any trial-related activities.
* Patients aged 18 years or older.
* Patients initiating injectable anticancer treatment (chemotherapy, immunotherapy, targeted therapies etc.).
* Patients with the capacity, personally (e.g., language and capacity to use the application), and in terms of infrastructure (internet access, possessing a smart phone etc.) to perform Cureety telemonitoring.
* Patient affiliated to an appropriate social security system

Non-inclusion criteria

* Exclusive oral cancer treatment
* Patient with dysphonia or difficulty communicating orally
* Patient benefiting from injectable cancer treatment as part of a clinical trial
* Inability to undergo trial monitoring for geographical, social or psychological reasons
* Any associated medical or psychological condition that could compromise the patient's ability to participate in the study
* Patient deprived of freedom or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Effectiveness of adding Cureety telemonitoring to usual care | 2 months
  Measured by number of outgoing calls to patients performing injectable anticancer treatments

CONTACTS AND LOCATIONS:
Overall Officials: Audrey FAVEYRIAL, MD, Principal Investigator — Centre François Baclesse
Locations (3):
- France (3):
  - Centre hospitalier de Bligny, Bligny
  - Centre François Baclesse, Caen
  - Centre de Radiothérapie et Oncologie Médicale d'Osny, Osny